CLINICAL TRIAL: NCT06608784
Title: Comparison Study of Electrocardiogram Indexes in Patients With Epilepsy, Patients With First Seizure and Normal Population
Status: Completed | Type: Observational
Sponsor: Mazandaran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Nasim Tabrizi, Associate Professor of Neurology, Mazandaran University of Medical Sciences
Other Study IDs: 15028; 15028 (Other: Mazandaran University of Medical Sciences)
Record Dates: First submitted 2024-09-13; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Patients With Epilepsy; Patients With First Seizure; Normal Population
Keywords: Electrocardiogram; Epilepsy; Seizure
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- Patients with epilepsy: Patients with epilepsy who experienced a recent generalized tonic-clonic seizure
  Interventions: Diagnostic Test: Electrocardiography
- Patients with first seizure: Patients who experienced a recent generalized tonic-clonic seizure without any previous history
  Interventions: Diagnostic Test: Electrocardiography
- Normal population: Participants without history of seizure or epilepsy
  Interventions: Diagnostic Test: Electrocardiography

INTERVENTIONS:
Diagnostic Test: Electrocardiography — 12-lead electrocardiography

SUMMARY:
According to recent advances in epileptic heart and sudden unexplained death in epilepsy, in this study the investigators aimed to compare ECG findings in patients with epilepsy, patients who had experienced their first seizure and patients without history of seizure.

ELIGIBILITY:
Inclusion Criteria for group 1:

* History of epilepsy for at least 2 years
* Taking antiseizure medications

Inclusion Criteria for group 2:

- Solid history of first seizure confirmed by a neurologist

Inclusion Criteria for group 3:

- No history of seizure

Exclusion Criteria:

* History of known cardiac disease or medical condition precipitating cardiac disease
* Electrolyte imbalance Taking medications with significant effect on ECG indexes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Three groups enrolled the study. The first group: Patients with epilepsy who experienced a generalized tonic-clonic seizure within 24 hours before admission.
  The second group: Patients who experienced a first time generalized tonic-clonic seizure within 24 hours before admission.
  The third group: Patients without a history of generalized tonic-clonic seizure.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-08-10 (Actual)

PRIMARY OUTCOMES:
Differences between ECG indexes in study groups | The ECG in group 1 and 2 was performed for patients who were admitted within 24 hours of seizure occurrence
  Analysis and comparing ECG indexes in study groups

CONTACTS AND LOCATIONS:
Locations (1):
- Mazandaran University of Medical Sciences, Sari, Mazandaran, Iran

IPD SHARING:
Plan to Share IPD: Yes
If needed based on request.
Supporting Information: Study Protocol